CLINICAL TRIAL: NCT06824519
Title: A Randomized, Blinded Phase I./II Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant
Brief Title: Clinical Trials of Quadrivalent Influenza Vaccine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LKM-2024-FIn-001
Record Dates: First submitted 2025-01-22; First posted 2025-02-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-02

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Phase I cohort 1 low-dose group (Experimental): 20 subjects aged 18-49 were enrolled and randomly assigned to the low-dose experimental group, and received one dose of the low-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (low dose)
- Phase I cohort 1 low-dose placebo group (Placebo Comparator): 10 subjects aged 18-49 were enrolled and randomly assigned to the low-dose placebo group, and received one dose of the low-dose placebo.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant placebo (low dose)
- Phase I cohort 2 high-dose group (Experimental): 20 subjects aged 18-49 were enrolled and randomly assigned to the high-dose experimental group, and received one dose of the high-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (high dose)
- Phase I cohort 2 high-dose placebo group (Placebo Comparator): 10 subjects aged 18-49 were enrolled and randomly assigned to the high-dose placebo group, and received one dose of the high-dose placebo.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant placebo (high dose)
- Phase I cohort 3 low-dose group (Experimental): 20 subjects aged 50 and above were enrolled and randomly assigned to the low-dose experimental group, and received one dose of the low-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (low dose)
- Phase I cohort 3 low-dose placebo group (Placebo Comparator): 10 subjects aged 50 and above were enrolled and randomly assigned to the low-dose placebo group, and received one dose of the low-dose placebo.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant placebo (low dose)
- Phase I cohort 4 high-dose group (Experimental): 20 subjects aged 50 and above were enrolled and randomly assigned to the high-dose experimental group, and received one dose of the high-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (high dose)
- Phase I cohort 4 high-dose placebo group (Placebo Comparator): 10 subjects aged 50 and above were enrolled and randomly assigned to the high-dose placebo group, and received one dose of the high-dose placebo.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant placebo (high dose)
- Phase II low-dose group (18-49 years old) (Experimental): 100 subjects aged 18-49 were enrolled and randomly assigned to the low-dose experimental group, and received one dose of the low-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (low dose)
- Phase II high-dose group (18-49 years old) (Experimental): 100 subjects aged 18-49 were enrolled and randomly assigned to the high-dose experimental group, and received one dose of the high-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (high dose)
- Phase II positive control group (18-49 years old) (Active Comparator): 50 subjects aged 18-49 were enrolled and randomly assigned to the positive control group, and received one dose of the positive control vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent
- Phase II low-dose group (50 years old and above) (Experimental): 100 subjects aged 50 and above were enrolled and randomly assigned to the low-dose experimental group, and received one dose of the low-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (low dose)
- Phase II high-dose group (50 years old and above) (Experimental): 100 subjects aged 50 and above were enrolled and randomly assigned to the high-dose experimental group, and received one dose of the high-dose experimental vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (high dose)
- Phase II positive control group (50 years old and above) (Active Comparator): 50 subjects aged 50 and above were enrolled and randomly assigned to the positive control group, and received one dose of the positive control vaccine.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent

INTERVENTIONS:
Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (low dose) — Inject 1 dose of low-dose vaccine
  Arms: Phase I cohort 1 low-dose group; Phase I cohort 3 low-dose group; Phase II low-dose group (18-49 years old); Phase II low-dose group (50 years old and above)
Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant placebo (low dose) — Inject 1 dose of low-dose placebo
  Arms: Phase I cohort 1 low-dose placebo group; Phase I cohort 3 low-dose placebo group
Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant (high dose) — Inject 1 dose of high-dose vaccine
  Arms: Phase I cohort 2 high-dose group; Phase I cohort 4 high-dose group; Phase II high-dose group (18-49 years old); Phase II high-dose group (50 years old and above)
Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant placebo (high dose) — Inject 1 dose of high-dose placebo
  Arms: Phase I cohort 2 high-dose placebo group; Phase I cohort 4 high-dose placebo group
Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent — Inject 1 dose of positive control vaccine
  Arms: Phase II positive control group (18-49 years old); Phase II positive control group (50 years old and above)

SUMMARY:
This clinical trial adopts a seamless design of phase I/II, conducted in two stages: phase I and phase II. Phase I is the age/dose ramp up stage, and phase II is the dose expansion stage.The purpose of this clinical trial is to evaluate the safety and tolerability of different doses of Influenza Vaccine (Split Virion), Inactivated, Quadrivalent, ZFA02 Adjuvant，explore the immunogenicity of the vaccine, and determine the appropriate dose for later clinical trials of this product.

DETAILED DESCRIPTION:
Overall design:

Adopting a randomized, blinded research design. This experiment adopts a seamless connection design of Phase I/II, conducted in two stages: Phase I and Phase II. Phase I is the age/dose escalation stage, and Phase II is the dose extension stage.

Age/dose escalation stage: A randomized, blinded, placebo-controlled study design was used. 120 subjects were enrolled in the study, in order of age from 18 to 49 years old to 50 years old and above, from low dose to high dose. They were divided into four cohorts, with 30 subjects in each cohort (including 20 who received high-dose or low-dose experimental vaccines and 10 who received placebo). The first 6 subjects in each cohort were assigned to be sentinel group, and the researchers reviewed the safety data of the sentinel group within 7 days after vaccination. After confirming safety (not meeting the criteria for suspending/terminating the trial), the remaining 24 subjects in the cohort were enrolled.

Dose expansion stage: A randomized, blinded, positive controlled study design was used. 500 subjects were enrolled, divided into two age groups: 18-49 years old and 50 years old and above. 250 subjects were enrolled in each age group and randomly divided into low-dose group, high-dose group, and positive control group according to a 2:2:1 ratio. The proportion of people aged 60 and above in the population aged 50 and above shall not be less than 80%, and the proportion of people aged 70 and above shall not be less than 30%.

ELIGIBILITY:
Inclusion Criteria:

1. When signing the informed consent form, be at least 18 years old and provide valid identification;
2. The subject is able to understand the procedures and methods of this clinical trial, has given sufficient informed consent, voluntarily participated, and signed an informed consent form by the subject themselves;
3. On the day of enrollment, axillary temperature was ≤ 37.0 ℃;
4. Female and male participants of childbearing age: agree to take effective contraceptive measures within 6 months after vaccination.

Exclusion Criteria:

1. The laboratory test indicators specified in the protocol are abnormal and clinically significant before vaccination (only for Phase I);
2. Have contracted influenza within the past 6 months prior to enrollment (confirmed by any clinical or microbiological method);
3. Previously or currently suffering from autoimmune or immunodeficiency diseases;
4. Previous history of severe allergies to any vaccine/drug or any component of the experimental vaccine, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, respiratory distress, angioneurotic edema, or individuals with an allergic constitution (such as allergies to two or more drugs, food, or pollen); History of severe allergy to eggs or egg protein;
5. Have received any influenza vaccine within the 6 months prior to enrollment, or plan to receive influenza vaccine other than the vaccine used in this trial during the trial period (before completing the immunization and collecting blood samples);
6. Within 30 days prior to enrollment, any investigational or unregistered products (drugs, vaccines, or devices) have been used, or are planned to be used during the trial period (except for the vaccine used in this trial) (before completing the immunization and collecting blood samples);
7. The interval between receiving attenuated live vaccines before enrollment is less than 30 days, and the interval between receiving other non live vaccines is less than 14 days;
8. Within the first 3 days of enrollment, have experienced acute illness or are in the acute phase of chronic illness;
9. Used antipyretic, analgesic, or anti allergic drugs within 3 days prior to enrollment;
10. Use immunoglobulin and/or any blood products within 3 months prior to enrollment, or plan to use them during the trial period (before completing immunization and collecting blood samples);
11. Long term use of immunosuppressants or other immunomodulatory drugs (defined as continuous use for more than 14 days) within the first 3 months of enrollment, such as a glucocorticoid dose of ≥ 0.5 mg/kg/day (inhalation and local steroid hormones are not restricted);
12. Absence of spleen, functional absence of spleen, and splenectomy caused by any condition;
13. Any obvious coagulation dysfunction or history of anticoagulant therapy;
14. History of epilepsy, encephalopathy, and malignant tumors;
15. Suffering from serious cardiovascular system diseases, serious hypertension with unstable drugs (systolic pressure ≥ 160mmHg and/or diastolic pressure ≥ 100mmHg), diabetes with serious complications and other serious chronic diseases;
16. Currently suffering from respiratory system diseases (including pneumonia, tuberculosis, severe asthma, chronic bronchitis, etc.), acute liver and kidney diseases (severe impairment of liver and kidney function), mental disorders (such as schizophrenia, depression, affective disorders, etc.), etc;
17. Women of childbearing age who are breastfeeding, pregnant, or have a positive urine pregnancy test before enrollment;
18. Plan to move out of the local area before the end of the study or plan to leave the local area for a long time during the study visit;
19. According to the researchers' judgment, the subjects have any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
AE occurren | within 30 days after vaccination
  Number and incidence of all adverse events
AESI occurrences | within 30 days after vaccination
  Number and incidence of all adverse events of special interest
SAE occurrences | within 12 months after vaccination
  Number and incidence of all serious adverse events
Serum alanine aminotransferase level | on the 4th day after vaccination
  All participants in Phase I were tested for alanine aminotransferase levels before and on the 4th day after vaccination
Serum aspartate transaminase level | on the 4th day after vaccination
  All participants in Phase I were tested for aspartate transaminase levels before and on the 4th day after vaccination
Serum total bilirubin level | on the 4th day after vaccination
  All participants in Phase I were tested for total bilirubin levels before and on the 4th day after vaccination
Serum white blood cell level | on the 4th day after vaccination
  All participants in Phase I were tested for white blood cell levels before and on the 4th day after vaccination
Serum platelet level | on the 4th day after vaccination
  All participants in Phase I were tested for platelet levels before and on the 4th day after vaccination
Serum hemoglobin level | on the 4th day after vaccination
  All participants in Phase I were tested for hemoglobin levels before and on the 4th day after vaccination
Urinary protein level in urine | on the 4th day after vaccination
  All participants in Phase I were tested for urinary protein levels in urine before and on the 4th day after vaccination
Urinary red blood cell level in urine | on the 4th day after vaccination
  All participants in Phase I were tested for urinary red blood cell levels in urine before and on the 4th day after vaccination
Serum antibody level | 30 days after vaccination
  Detect the levels of hemagglutination inhibition (HI) antibodies against influenza viruses H1N1, H3N2, and type B (B/Victoria and B/Yamagata).

CONTACTS AND LOCATIONS:
Overall Officials: Fei Jin, Principal Investigator — Hebei Province Centers for Disease Control and Prevention
Locations (1):
- Hebei Province Centers for Disease Control and Prevention, Shijiazhuang, Hebei, China